CLINICAL TRIAL: NCT00143377
Title: A Global Phase IV, Double-Blind, Placebo-Controlled, Randomized Trial To Evaluate The Effectiveness Of Detrusitol Sr 4mg On Patient's Perception Of Bladder Condition (PPBC).
Brief Title: Study to Determine The Effectiveness Of Detrusitol In Patients Diagnosed With OAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Pfizer (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121122
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

INTERVENTIONS:
Drug: tolterodine SR, overactive bladder

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Detrusitol (tolterodine tartrate) SR, 4 mg once daily, on patient's perception of the symptoms of overactive bladder and which of these bothersome symptoms are improved with treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older patients suffering from OAB symptoms (urinary frequency of at least 8 micturitions per 24h, urinary urgency and at least 3 urge urinary incontinence episodes within 3 days), confirmed by a micturition bladder diary.

Exclusion Criteria:

* Other than urge incontinence
* History of prostate/uterine or other female organ cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-09; Study Completion 2005-10

PRIMARY OUTCOMES:
Patient Perception of Bladder Condition at 12 weeks of treatment compared to placebo.

SECONDARY OUTCOMES:
Other safety and efficacy measures at 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Herschorn S, Heesakkers J, Castro-Diaz D, Wang JT, Brodsky M, Guan Z; Disease Management Study Team. Effects of tolterodine extended release on patient perception of bladder condition and overactive bladder symptoms*. Curr Med Res Opin. 2008 Dec;24(12):3513-21. doi: 10.1185/03007990802537122. PMID 19032133